CLINICAL TRIAL: NCT05368597
Title: Comparison of Percutaneous Coronary Intervention in Native Arteries Versus Bypass Grafts in Patients With Prior Coronary Artery Bypass Grafting
Brief Title: CompArison of PCI in NaTive Arteries Versus ByPAss Grafts In PatieNts With Prior CABG (CAPTAIN)
Status: Completed | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Yujie Zhou, Clinical Professor, Beijing Anzhen Hospital
Other Study IDs: CAPTAIN
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery bypass grafting; percutaneous coronary intervention; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Native vessel PCI: Native vessel PCI, which choose native coronary artery as the target vessel
  Interventions: Procedure: PCI in native vessel or in bypass graft
- Bypass graft PCI: Bypass graft PCI, which choose the graft vessel as the target vessel
  Interventions: Procedure: PCI in native vessel or in bypass graft

INTERVENTIONS:
Procedure: PCI in native vessel or in bypass graft — Native vessel PCI,which choose native coronary artery as the target vessel, while the bypass graft PCI choose graft vessel as the target vessel.

SUMMARY:
Coronary atherosclerotic heart disease (CAD) has been considered the leading cause of death in both developed and developing countries. Coronary artery bypass grafting (CABG) is a major therapy of CAD in the world, mainly used for patients with left main disease, multi-vessel complex disease, stent implantation failure, heart failure and diabetes.

Studies have demonstrated that significant angiographic defects up to 12% of grafts, which was observed by immediate coronary angiography after CABG. Despite secondary prevention were performed in patients after CABG, the early failure rate at 1 year is higher, up to 15-20%, the 10-year patency rate of internal mammary artery graft is 85%, and the 10-year patency rate of saphenous vein graft is only 61%, and 10-20% of patients require revascularization within 10 years after CABG.

Patients with failed grafts usually have a higher surgical risk and the morality of repeat CABG is 2-4 times higher than primary surgery. Because of the poor clinical prognosis of patients undergoing repeat CABG, PCI is the preferred treatment strategy for revascularization in patients with previous CABG. In patients with previous CABG, approximately 75% of PCI target vessels are native vessels.

Compared with native vessel PCI, bypass graft PCI has a higher rate of short- and long-term major adverse events, including more than double the in-hospital mortality rate. Some studies support the above view，but others denied. Therefore, the primary study mainly to explore the effect of native vessel PCI or graft PCI on the prognosis of patients with previous CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients received first percutaneous coronary intervention in native arteries or in bypass grafts after coronary artery bypass grafting

Exclusion Criteria:

* Patients who missed follow-up data were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Coronary artery disease patients received first percutaneous coronary intervention in native arteries or in bypass grafts after coronary artery bypass grafting
Sampling Method: Non-Probability Sample
Enrollment: 1491 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular event (MACE) | about 10 years after PCI
  A composite of all-cause death, non-fatal stroke, non-fatal myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Wang, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No